CLINICAL TRIAL: NCT00460005
Title: A Multicenter Study to Determine the Clinical Characteristics of the Temporal Aspects of Migraine in a Canadian Population: Clinical Study Of Migraine Evolution (C-SOME)
Brief Title: Clinical Study Of Migraine Evolution
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Other Study IDs: S2W106188
Record Dates: First submitted 2007-04-12; First posted 2007-04-13 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Migraine Headache
Keywords: Migraine; headache; observational
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Understanding the speed at which migraine headaches develop is of importance to patients. Determining the proportions in which different headache pain build-up occurs, may provide health care practitioners with valuable information with which to prescribe the most appropriate treatment. Patients who experience a slow pain build-up may gain more benefit from medications which have a slow onset of effect, high tolerability and long action. Conversely, medications with a rapid onset of effect may be of greater benefit to patients who experience rapid onset of migraine pain.

ELIGIBILITY:
Inclusion Criteria:

* Subject is outpatient.
* Subject has a diagnosis of migraine with/without aura according to IHS criteria, of at least 1 years duration.
* Subject is able to comprehend the study procedures and to comply with study requirements.

Exclusion Criteria:

* Subject has other chronic pain condition(s) not associated with migraine
* Subject is unable to understand the schedule/questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, M.D., Study Director — GlaxoSmithKline
Locations (10):
- Canada (10):
  - GSK Clinical Trials Call Centre, Calgary, Alberta
  - GSK Clinical Trials Call Centre, Richmond, British Columbia
  - GSK Clinical Trials Call Centre, Vancouver, British Columbia
  - GSK Clinical Trials Call Centre, Saint John, New Brunswick
  - GSK Clinical Trials Call Centre, Halifax, Nova Scotia
  - GSK Clinical Trials Call Centre, Hamilton, Ontario
  - GSK Clinical Trials Call Centre, Toronto, Ontario
  - GSK Clinical Trials Call Centre, Unionville, Ontario
  - GSK Clinical Trials Call Centre, Longueuil, Quebec
  - GSK Clinical Trials Call Centre, Montreal, Quebec